CLINICAL TRIAL: NCT00935935
Title: A Pilot Study on the Immunopathogenesis of Bone Disease in Older HIV-infected Adults
Brief Title: Study of Bone Disease in Older HIV-infected Adults
Status: Completed | Type: Observational
Sponsor: Ruth M. Rothstein CORE Center (Other)
Collaborators: Rush University Medical Center (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, oluwatoyin M. Adeyemi, principal investigator, Ruth M. Rothstein CORE Center
Other Study IDs: Bone2009
Record Dates: First submitted 2009-07-08; First posted 2009-07-09 (Estimated); Last update posted 2012-08-03 (Estimated); Status verified 2012-08

CONDITIONS: Osteopenia; Osteoporosis; HIV Infection; Aging; HIV Infections
Keywords: Treatment experienced
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV older than 50 years

SUMMARY:
This study will look to see if there are changes in the blood cells that are associated with bone disease and sort out effects that are due to the HIV virus itself, the medications and see if faster aging occurs in the cells of HIV infected persons. Bone disease will be measured by a special X-ray called a DEXA scan. A DEXA scan is used by doctors to see if someone has normal bone mass for their age or if there is thinning of the bones.

The purposes of this study are:

* to learn how common bone disease is in HIV infected patients over the age of 50 years that receive their care at the CORE Center
* to see what are the common causes of bone disease in older HIV infected persons
* to see if there are differences in blood cells and levels of cytokines in patients who do or do not have bone disease, as this may help researchers determine the cause of bone disease.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection documented by ELISA and confirmed by western blot
* Treatment with antiretroviral drugs for at least 12 months
* Age 50-70 years
* CD4 count > 350 cells/mm3 for at least 6 months
* HIV-RNA undetectable (< 75 copies/ml for at least 6 months)

Exclusion Criteria:

* Known bone disease (primary or metastatic malignancy, osteomalacia)
* Treatment for bone disease (bisphosphonates, calcitonin, strontium, sodium fluoride, synthetic PTH, or high-dose vitamin D [> 800 IU daily]).

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 HIV-infected adults, age 50 years or older, on HAART with undetectable viral loads, who are randomly sampled from 6 strata defined by ethnicity (Black:White:Hispanic; 2:1:1) and sex (male:female; 1:1).
  100 HIV+ adults, age ≥ 50 yr (50 ♂, 50 ♀; 50 AA, 25 W, 25 H).
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assess the associations between outcome (bone density) and predictors (markers of inflammation and immune activation) using continuous variables | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Oluwatoyin Adeyemi, MD, Principal Investigator — Ruth M. Rothstein CORE Center
Locations (1):
- Ruth M Rothstein CORE Center, Chicago, Illinois, United States